CLINICAL TRIAL: NCT05724680
Title: A Randomized Controlled Trial of the Effectiveness of Cognitive Behavior Therapy for Major Depression in Bangladesh
Brief Title: Effectiveness of Cognitive Behavior Therapy for Persons With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajshahi University (Other)
Collaborators: University Grants Commission (Other)
Responsible Party: Principal Investigator, Dr. Jesan Ara, Associate Professor, Rajshahi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-PhD/2017/1985
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): cognitive behavior therapy
  * one session per week
  * six to eight session
  Interventions: Other: cognitive behavior therapy
- Wait list control group (Other): * waitlist control group
  * offer CBT after completing data collection.
  Interventions: Other: cognitive behavior therapy

INTERVENTIONS:
Other: cognitive behavior therapy — Psycho-therapeutic intervention

SUMMARY:
This was a randomized controlled clinical trial (RCT) carried out in three different hospitals in Dhaka city, Bangladesh.

DETAILED DESCRIPTION:
This was a randomized controlled trial, conducted to determine the effectiveness of CBT for depression delivered by trained therapists with an adapted Bengali CBT (BaCBT) manual, as compared to a control group. The main objective of the current study was to examine the efficacy of CBT for persons with major depression in Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Major Depression
* Must be able to take therapeutic session

Exclusion Criteria:

* active suicidal ideation
* a co-morbid serious health condition
* with psychotic features
* currently on medication for depression
* with an intellectual disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Depression Scale | change from baseline to day 42, a separate outcome from day 42 to day 72
  Depression Scale to measure depression. The total scale scores range from 30 to 150. Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Change in Anxiety Scale | change from baseline to day 42, a separate outcome from day 42 to day 72
  Anxiety Scale, the possible range of scores from 0 to 144 and Higher scores mean worse outcomes.
Change in General Health Questionnaire-28 | change from baseline to day 42, a separate outcome from day 42 to day 72
  General Health Questionnaire-28, range of scores from 0 to 84, and Higher scores mean worse outcomes.
Change in Beck Scale for Suicidal Ideation | change from baseline to day 42, a separate outcome from day 42 to day 72
  Beck Scale for Suicidal Ideation, range of scores from 0 to 42, and Higher scores mean worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Jesan ara, Rajshahi, Rajshahi Division, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
Analysis of data will be shared through research publications.